CLINICAL TRIAL: NCT02015390
Title: The Comparative Efficacy of the Masquelet Versus Titanium Mesh Cage Reconstruction Techniques for the Treatment of Large Long Bone Deficiencies
Brief Title: Comparative Efficacy of the Masquelet Versus Titanium Mesh Cage Techniques for the Treatment of Large Long Bone Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-100; DoD OR120128 (Other: US Department of Defense PRORP)
Record Dates: First submitted 2013-05-29; First posted 2013-12-19 (Estimated); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Segmental Long Bone Defects
Keywords: bone defects; iatrogenic resection; titanium mesh cage; biomembrane; Masquelet technique
MeSH Terms: interventions — Transplantation, Homologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Masquelet defect reconstruction (Active Comparator): The Masquelet defect reconstruction is a two-stage technique for the treatment of large segmental bone defects that involves the induction of a biomembrane about a poly(methylmethacrylate)(PMMA) cement spacer within the defect and, following cement removal, autogenous bone grafting (harvested using Reamer-Irrigator-Aspirator) or allogeneic bone graft is used to pack the defect while preserving the biomembrane. The typical time interval between the two stages is 6-8 weeks. The biomembrane not only assists in retaining the bone graft, but serves as a rich source of vascular supply and growth factors which constitute an excellent biological milieu for the graft to consolidate and heal the defect.
  Interventions: Procedure: Autogenous RIA bone grafting; Procedure: Allogeneic bone grafting
- Titanium cage reconstruction (Active Comparator): The cylindrical titanium mesh cage technique is a single-stage surgical procedure that immediately restores limb anatomy and alignment, and provides limb stability sufficient enough for early, unrestricted mobilization while permitting bone and soft tissue healing. It involves the implantation of a fenestrated cylindrical titanium mesh cage packed with autogenous bone graft (harvested using Reamer-Irrigator-Aspirator) or with allogeneic bone graft.
  Interventions: Procedure: Autogenous RIA bone grafting; Procedure: Allogeneic bone grafting

INTERVENTIONS:
Procedure: Autogenous RIA bone grafting — After aseptic defect and adequate soft tissue coverage have been achieved, the defect reconstruction technique will include autogenous bone grafting harvesting using Reamer-Irrigator-Aspirator (RIA) and packing it within the defect.
  Other Names: RIA grafting
Procedure: Allogeneic bone grafting — After aseptic defect and adequate soft tissue coverage have been achieved, the defect reconstruction technique will include defect packing with allogeneic bone graft croutons combined with demineralized bone matrix (DBM).
  Other Names: Allograft

SUMMARY:
The United States Department of Defense (DoD) is funding exciting new research at the University of Texas Medical Branch (UTMB) Department of Orthopaedic Surgery and Rehabilitation that can be a major improvement in the treatment of extremity trauma involving segmental bone loss. These devastating injuries occur frequently in both civilians and the military. They typically result from motor vehicle accidents, high-energy fractures, gunshot injuries, and blast injuries, but also from the surgical removal of a bone segment because of infection or tumor. Despite many modern medical advances in this area, bone healing that can adequately replace bone loss and restore pre-injury limb function is extremely difficult to achieve. Existing standard treatment procedures are exceedingly complicated, require highly specialized equipment and clinical skills, and usually require many surgical procedures over many months or years. Despite these effort and costs, major complications usually occur with all the standard treatment options, the patient's ability to return to an acceptable functional status is typically low, and, therefore, many of these patients have their limbs amputated.

The UTMB Department of Orthopaedic Surgery and Rehabilitation will conduct a DoD-funded clinical trial to determine and compare the advantages of two new and innovative surgical bone defect treatment techniques that can be significantly more effective for wounded warriors or civilian patients and with these conditions. One treatment method, called "the Masquelet Technique", involves two-stage surgery: the first one to create a biomembrane around the defect by applying a cement spacer, and then the second one for cement spacer removal and defect bone grafting. The other method, developed by UTMB physicians, is "the Cage Technique" and it comprises one-stage surgery in which a special hollow, fenestrated, titanium cage filled with bone graft is implanted in the defect. Initial clinical experience with both of these techniques has been very promising, but to date, there has been no prospective clinical study comparing the two new methods of defect treatment. Identifying an optimal surgical bone defect reconstructive technique would significantly improve the clinical outcomes of patients with these challenging conditions.

DETAILED DESCRIPTION:
Background: Segmental long bone defects remain a formidable treatment challenge. All the existing standard treatment options have major limitations and often culminate in limb amputation or permanent functional deficits. We developed a novel, one-stage alternative treatment for segmental bone loss that utilizes the cylindrical titanium mesh cage (CTMC) in combination with bone graft, and have established its clinical merits in an initial clinical series. Shortly thereafter, Masquelet reported another new defect reconstruction technique that involves two-stage approach: first inducing biomembrane formation with a cement spacer, and subsequent spacer removal and bone grafting. Both the Masquelet and the CTMC techniques are based on the principle of graft containment to render optimal potential for graft to heal the defect; however, they differ in primary biological versus biomechanical functions provided by the containment. The Masquelet biomembrane containment, being a rich source of vascular supply and growth factors, creates an excellent biological milieu for graft, but requires an additional surgery and is associated with prolonged protected weight bearing until graft consolidation occurs. Conversely, the benefit of the CTMC technique is primarily the biomechanical support it provides for graft and the reconstructed extremity, thereby permitting immediate functional restoration without mobility or weight bearing restrictions during the bone healing process. Although both Masquelet and the CTMC techniques have been effective in the treatment of large segmental bone defects, there is no prospective, well-controlled study comparing their therapeutic efficacies for specific clinical indications.

Objective: Determining the clinical efficacy and cost-effectiveness of the Masquelet (Arm I) versus the CTMC technique (Arm II) in combination with reamer-irrigator-aspirator (RIA) harvested autograft (Option A) or allograft-demineralized bone matrix (DBM) composite (Option II) in the treatment of segmental long bone deficiencies.

Specific Aims: 1) Establish the effects of the specific patient and bone defect characteristics on the treatment outcome; 2) Determine and compare clinical efficacies of the reconstruction techniques (Arm I vs Arm II); 3) Establish the merits of using specific graft type (Option A vs Option B) within and across each study arms; 3) Develop a quantitative predictive model to improve clinical decision making, and 4) Assess and compare the cost-effectiveness and resource expenditures incurred by the specific treatment selection.

Study Design: Single-center, multi-site, two-arm, randomized clinical trial. Thirty patients with segmental bone deficiency as a result of trauma, gunshot, iatrogenic resection due to infection, nonunion, or neoplasm will be enrolled and randomized to receive either the Masquelet (Arm I) or the CTMC as definitive defect treatment (Arm II). Bone graft selection will include either RIA-harvested autograft (Option A) or allograft croutons-DBM composite (Option B). Patients will be followed up to18 months. The data collected will include routine patient baseline information, systemic and extremity injury characteristics, bone defect characteristics, pre- and post-operative clinical examinations and imaging, validated functional outcomes measures, and associated cost expenditure. Descriptive statistics will be used to analyze and compare the results specifically related to the rate of defect healing and functional recovery. Paired t-test will be used to test the effects of the defect reconstruction option on the outcome measures. Analysis of covariance will be used for pair-wise comparison between the arms and within/across each bone graft option. Multiple models will be used to produce an accurate predictive model which accounts for possible morbidities and interactions. Derived from the joint distribution of costs and effects, cost-effectiveness acceptability curves will be established and compared for the study arms.

Military Relevance: Many combat injuries involve extremity trauma with segmental bone loss, and the extent to which they can be successfully treated impacts the function and quality of life of the wounded warrior. The Masquelet and the CTMC been developed as innovative, biologically-sound defect reconstructive techniques to address the complexity of therapeutic concerns associated with these conditions (ie, immediate restoration of limb alignment/stability, early motion, weight bearing). The proposed trial aims to compare the efficacy of these techniques to identify the one that can be instantly adopted and applied by military surgeons.

ELIGIBILITY:
Inclusion Criteria:

Presence of an extremity long bone (femur, tibia, humerus, ulna, radius) segmental defect requiring surgical reconstruction with at least one of the following etiologies:

* traumatic segmental bone defect that warrants surgical reconstruction;
* acquired bony nonunion (not congenital) treatable by segmental resection and reconstruction;
* local osteomyelitis (dormant or active) treatable by segmental bone resection and reconstruction;
* localized, nonmalignant tumor with involvement of bone diaphysis treatable by segmental bone resection and reconstruction.

Exclusion Criteria:

* Non-segmental defects (eg, defect in continuity involving only single cortex);
* Inability or contraindications to achieve stabilization with an intramedullary (IM) nail;
* Insufficient defect size (humerus defects <5 cm; femur or tibia defect <2 cm in length);
* Extremity unsuitable for salvage;
* Patients with inadequate neuro-vascular status;
* Defect and/or soft tissue status ineligible for surgical reconstruction;
* Ipsilateral extremity defect (eg, tibia and femur ipsilateral defects);
* Skeletal immaturity (open growth plate and/or age <18 years);
* Known allergic reaction to titanium implants;
* Disseminated osteomyelitis throughout the bone;
* Active systemic infection at time of surgery;
* Congenital / genetic etiology of nonunion (congenital pseudoarthrosis, osteogenesis imperfecta, etc.);
* Women who are pregnant or nursing;
* Women who intend to become pregnant during the study followup (ie, 2 years);
* Disseminated and/or nonresectable malignant tumor involving bone;
* Patients with active compartment syndrome;
* Prisoners;
* Patients considered as non-compliant with medical and follow up care;
* Patients using narcotics, abusing prescription drugs (within last 2 years);
* Patients with alcohol abuse;
* Patients deemed incapable of following instructions pertaining to post operative care due to mental or medical condition;
* Patients deemed ineligible due to medico-social concerns.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew Gugala, MD,PhD, Principal Investigator — University o Texas Medical Branch in Galveston, Texas; Ronald W Lindsey, MD, Principal Investigator — University o Texas Medical Branch in Galveston, Texas
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 8 screen failures
Groups:
- Masquelet Defect Reconstruction: The Masquelet defect reconstruction is a two-stage technique for the treatment of large segmental bone defects that involves the induction of a biomembrane using a poly(methylmethacrylate)(PMMA) cement spacer followed by cement removal and bone grafting of the defect while preserving the biomembrane. The biomembrane not only assists in retaining the bone graft, but serves as a rich source of vascular supply and growth factors which constitute an excellent biological milieu for the graft to consolidate and heal the defect.
  The first stage of the Masquelet defect reconstruction involves creating a biomembrane with a PMMA spacer; whereas the second stage performed 6-8 weeks later involves the spacer removal and packing the defect enclosed with the biomembrane with autogenous (RIA) or allogeneic bone graft. The biomembrane serves as a biological enclosure for the graft, provides vascular supply and growth factors, thereby creating an excellent milieu for the graft to consolidate.
- Titanium Cage Reconstruction: The cylindrical titanium mesh cage technique is a single-stage surgical procedure that immediately restores limb anatomy and alignment, and provides limb stability sufficient enough for early, unrestricted mobilization while permitting bone and soft tissue healing. It involves the implantation of a fenestrated cylindrical titanium mesh cage packed with autogenous bone graft (harvested using Reamer-Irrigator-Aspirator) or with allogeneic bone graft.
  After aseptic defect and soft tissue bed is achieved, the titanium cage reconstruction procedure involves the implantation of a fenestrated cylindrical titanium cage packed with simultaneously harvested autogenous bone graft using RIA or with allogeneic bone graft. The decision about the graft option is left for the treating physician, following the discussion with the patient. The cage provide a biomechanical enclosure for the graft, allows the graft to be loaded, and, thereby consolidate and heal the defect.
Period: Overall Study
Arm/Group | Masquelet Defect Reconstruction | Titanium Cage Reconstruction
Started | 9 | 7
Completed | 8 | 3
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 0 | 3
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: 16 patients in both arms with demographic characteristics as outlined below
Groups:
- Total: Total of all reporting groups
Arm/Group | Masquelet Defect Reconstruction | Titanium Cage Reconstruction | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Full Range); unit: years] | 53.56 [34 to 73] | 46.43 [38 to 59] | 50.43 [24 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Defect Healing - Plain Radiography
Description: Biplanar radiography to demonstrate adequate hardware placement and defect alignment in all patients in the Masquelet and Cage trial arms.
Time Frame: 2 weeks postop
Population: 2 week radiographic imaging
Measure: Count of Participants; unit: Participants
Arm/Group | Masquelet Defect Reconstruction | Titanium Cage Reconstruction
Number analyzed (Participants) | 9 | 7
Participants | 9 | 7

2. Primary Outcome: Number of Participants With Defect Healing - Plain Radiography
Description: Biplanar radiography to demonstrate defect and graft alignment in all patients in the Masquelet and Cage trial arms.
Time Frame: 6 weeks postop
Population: 6 week radiographic imaging
Measure: Count of Participants; unit: Participants
Groups:
- Titanium Cage Reconstruction: The cylindrical titanium mesh cage technique is a single-stage surgical procedure that immediately restores limb anatomy and alignment, and provides limb stability sufficient enough for early, unrestricted mobilization while permitting bone and soft tissue healing. It involves the implantation of a fenestrated cylindrical titanium mesh cage packed with autogenous bone graft (harvested using Reamer-Irrigator-Aspirator) or with allogeneic bone graft.
  After aseptic defect and soft tissue bed is achieved, the titanium cage reconstruction procedure involves the implantation of a fenestrated cylindrical titanium cage packed with simultaneously harvested autogenous bone graft using RIA or with allogeneic bone graft. The decision about the graft option is left for the treating physician, following the discussion with the patient. The cage provides a biomechanical enclosure for the graft, allows the graft to be loaded, and, thereby consolidate and heal the defect.
Arm/Group | Masquelet Defect Reconstruction | Titanium Cage Reconstruction
Number analyzed (Participants) | 9 | 3
Participants | 9 | 3

3. Primary Outcome: Number of Participants With Defect Healing - Plain Radiography
Description: Radiographic assessment to demonstrate the adequate bony alignment and hardware placements for all patients in the Masquelet and Cage trial arms maintained upon patients' active weightbearing.
Time Frame: 3 months postop
Population: 3 month radiographic imaging
Measure: Count of Participants; unit: Participants
Arm/Group | Masquelet Defect Reconstruction | Titanium Cage Reconstruction
Number analyzed (Participants) | 8 | 3
Participants | 8 | 3

4. Primary Outcome: Number of Participants With Defect Healing - Plain Radiography
Description: Radiographic biplanar determination of bone defect healing progression.
Time Frame: 6 months postop
Population: 6 month radiographic imaging
Measure: Count of Participants; unit: Participants
Arm/Group | Masquelet Defect Reconstruction | Titanium Cage Reconstruction
Number analyzed (Participants) | 8 | 3
Participants | 8 | 3

5. Primary Outcome: Number of Participants With Defect Healing - Plain Radiography
Description: Radiographic imaging to demonstrate bone graft consolidation and callus formation in the patients with the Masquelet reconstruction and cage techniques.
Time Frame: 12 months postop
Population: 12 month radiographic imaging
Measure: Count of Participants; unit: Participants
Arm/Group | Masquelet Defect Reconstruction | Titanium Cage Reconstruction
Number analyzed (Participants) | 8 | 3
Participants | 8 | 3

6. Primary Outcome: Number of Participants With Defect Healing - Plain Radiography
Description: Radiographic biplanar determination of bone defect healing to demonstrate bone graft consolidation and defect healing in all Masquelet- and Cage-treated patients who completed the trial.
Time Frame: 18 months postop
Population: 18 month radiographic imaging
Measure: Count of Participants; unit: Participants
Arm/Group | Masquelet Defect Reconstruction | Titanium Cage Reconstruction
Number analyzed (Participants) | 8 | 3
Participants | 8 | 3

7. Primary Outcome: Number of Participants With Defect Healing - Computed Tomography
Description: Radiographic spatial determination of bone defect healing
Time Frame: 12 months postop
Population: 12 month CT imaging
Measure: Count of Participants; unit: Participants
Arm/Group | Masquelet Defect Reconstruction | Titanium Cage Reconstruction
Number analyzed (Participants) | 8 | 3
Participants | 8 | 3

8. Primary Outcome: Number of Participants With Defect Healing - Computed Tomography
Description: Radiographic spatial determination of bone defect healing
Time Frame: 18 months postop
Population: 18 month CT imaging
Measure: Count of Participants; unit: Participants
Arm/Group | Masquelet Defect Reconstruction | Titanium Cage Reconstruction
Number analyzed (Participants) | 8 | 3
Participants | 8 | 3

9. Secondary Outcome: Pain Assessment: Brief Pain Inventory
Description: Brief Pain Inventory
Time Frame: 2 weeks postop
Reporting Status: Not Posted

10. Secondary Outcome: Pain Assessment: Brief Pain Inventory
Description: Brief Pain Inventory
Time Frame: 6 weeks postop
Reporting Status: Not Posted

11. Secondary Outcome: Pain Assessment: Brief Pain Inventory
Description: Brief Pain Inventory
Time Frame: 3 months postop
Reporting Status: Not Posted

12. Secondary Outcome: Pain Assessment: Brief Pain Inventory
Description: The patients in both the Masquelet and Cage trial arms demonstrated most significant improvement in Brief Pain Inventory scores at 12 month followup. No statistical differences were observed in pain score among the patients from both trial arms.
Time Frame: 6 months postop
Reporting Status: Not Posted

13. Secondary Outcome: Pain Assessment: Brief Pain Inventory
Description: The trial patients in both Masquelet and Cage arms demonstrated continued improvements in pains score at 12 months followup. No significant difference in pains core were noted between the trial arms.
Time Frame: 12 months postop
Reporting Status: Not Posted

14. Secondary Outcome: Pain Assessment: Brief Pain Inventory
Description: Brief Pain Inventory
Time Frame: 18 months postop
Reporting Status: Not Posted

15. Secondary Outcome: Overall Functional Outcome Score
Description: Short-Form 36
Time Frame: 2 weeks postop
Reporting Status: Not Posted

16. Secondary Outcome: Overall Functional Outcome Score
Description: Short-Form 36
Time Frame: 6 weeks postop
Reporting Status: Not Posted

17. Secondary Outcome: Overall Functional Outcome Score
Description: Short-Form 36
Time Frame: 3 months postop
Reporting Status: Not Posted

18. Secondary Outcome: Overall Functional Outcome Score
Description: Short-Form 36
Time Frame: 6 months postop
Reporting Status: Not Posted

19. Secondary Outcome: Overall Functional Outcome Score
Description: Short-Form 36
Time Frame: 12 months postop
Reporting Status: Not Posted

20. Secondary Outcome: Overall Functional Outcome Score
Description: Among patients who completed the trial for both the Masquelet and Cage arms, SF-36 demonstrated an overall progressive improvement in the score comportment, such as in Physical function (PF); Mental health (MH); Social function (SC); Bodily pain (BP); Change in health (CH); Vitality (VT); Role limitation - physical (RLP); Role limitation - mental (RLM); Health perception (HP). The most apparent improvements were observed in the Physical function (PF); Mental health (MH); Social function (SC); Bodily pain (BP); Change in health (CH); Vitality (VT) and Health perception (HP). No statistical difference were noted in overall SF-36 scores between the trail arms.
Time Frame: 18 months postop
Reporting Status: Not Posted

21. Secondary Outcome: Extremity-Specific Outcome Score
Description: Lower Limb Core Scale or Short Form the Arm, Shoulder, and Hand
Time Frame: 2 weeks postop
Reporting Status: Not Posted

22. Secondary Outcome: Extremity-Specific Outcome Score
Description: Lower Limb Core Scale or Short Form the Arm, Shoulder, and Hand
Time Frame: 6 weeks postop
Reporting Status: Not Posted

23. Secondary Outcome: Extremity-Specific Outcome Score
Description: Lower Limb Core Scale or Short Form the Arm, Shoulder, and Hand
Time Frame: 3 months postop
Reporting Status: Not Posted

24. Secondary Outcome: Extremity-Specific Outcome Score
Description: Lower Limb Core Scale or Short Form the Arm, Shoulder, and Hand
Time Frame: 6 months postop
Reporting Status: Not Posted

25. Secondary Outcome: Extremity-Specific Outcome Score
Description: Lower Limb Core Scale or Short Form the Arm, Shoulder, and Hand
Time Frame: 12 months postop
Reporting Status: Not Posted

26. Secondary Outcome: Extremity-Specific Outcome Score
Description: Lower Limb Core Scale or Short Form the Arm, Shoulder, and Hand
Time Frame: 18 months postop
Reporting Status: Not Posted

27. Secondary Outcome: Change in Quality of Life: Quality-Adjusted Life-Year
Description: An improvement in mean Quality Adjusted Life Years (QALY) calculated from the subjective pain questionnaire throughout the trial followup as a result of bone defect treatment for patients in the Masquelet Arm versus the Cage Arm. QALY values ranged from 0 to 1 referring to death and perfect health, respectively. There was apparent improvement in QALY at 6 month and 12 month post treatment for both trial arm patients compared to the preperative QALY scores. No statistically significant difference at any time point of the followup between the trial arms were noted.
Time Frame: from 2 weeks postop to 18 months postop
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Masquelet Defect Reconstruction | Titanium Cage Reconstruction
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 3/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Masquelet Defect Reconstruction (N=8) | Titanium Cage Reconstruction (N=7)
6 months post reconstructive surgery (Infections and infestations) | 0 (0) | 1 (1) — A 48-old male patients randomized to the Cage Arm for the treatment of his 5-cm-long midshaft tibial bone defect, presented to the clinic at 6-months post reconstructive surgery with infected draining wound and defect infection.
3 weeks post reconstructive surgery (Infections and infestations) | 0 (0) | 1 (1) — A 36-year-old female with a infected tibia nonunion treated with the Cage Technique and allograft developed wound dehiscence and defects infection which resulted from noncompliance with antibiotic therapy and intravenous illicit drug abuse.
18 months post reconstructive surgery (Infections and infestations) | 0 (0) | 1 (1) — A 47-year-old female who received the Cage reconstruction for a 6.5-cm midshaft humerus defect presented with infection 3 days before the final 18-month follow-up. Patient was reported as noncompliant with positive illegal drug amphetamine in blood.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT02015390/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT02015390/SAP_001.pdf